CLINICAL TRIAL: NCT07013981
Title: The Synchronized Trial on Expectant Mothers With Depressive Symptoms by Omega-3 PUFAs (SYNCHRO)in Tokyo: Open Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Science and Technology Council, Taiwan (Other Government)
Collaborators: Japanese Society for the Promotion of Science (Other); University of Toyama (Other); Chiba University (Other)
Responsible Party: Principal Investigator, Kuan-Pin, Professor, National Science and Technology Council, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH102-REC1-060
Record Dates: First submitted 2022-10-07; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression | interventions — Docosahexaenoic Acids; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 polyunsaturated fatty acids (Experimental): 1200mg EPA and 600mg DHA daily
  Interventions: Dietary Supplement: Omega-3 polyunsaturated fatty acids
- Placebo Comparator (Placebo Comparator): 320 mg olive oil and 9.9 mg omega-3 PUFAs
  Interventions: Dietary Supplement: Omega-3 polyunsaturated fatty acids

INTERVENTIONS:
Dietary Supplement: Omega-3 polyunsaturated fatty acids
  Other Names: 1200mg EPA and 600mg DHA daily
  Arms: Omega-3 polyunsaturated fatty acids
Dietary Supplement: Omega-3 polyunsaturated fatty acids
  Other Names: 320 mg olive oil and 9.9 mg omega-3 PUFAs
  Arms: Placebo Comparator

SUMMARY:
The present study aims to examine the efficacy and safety of omega-3 polyunsaturated fatty acids for pregnant women with depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. pregnant women aged 20 years or older.
2. between 12-24 weeks gestation.
3. a Japanese conversational ability to understand the scope of the present trial.
4. planned to return to the hospital for checkup at 4-6 weeks after childbirth.
5. an Edinburgh Postnatal Depression Scale (EPDS) score is 9 or more.
6. to have good physical health judged by obstetricians.

Exclusion Criteria:

1. history and current suspicion of psychosis or bipolar I disorder or substance-related disorder or eating disorder or personality disorder.
2. the item of EPDS concerning suicide ideation is 2 or more.
3. other serious psychiatric symptoms such as self-harm behavior or in need of rapid psychiatric treatment.
4. difficult to expect a normal birth (ex: fetal malformation etc.).
5. having a history of bleeding disorder such as von Willebrand's Disease.
6. regular treatment with aspirin or warfarin within the last 3 months.
7. a smoking habit of ≥40 cigarettes per day.
8. regular treatment with ethyl icosapentate or regular consumption of omega- 3 PUFA supplements within the last 3 months.
9. a habit of eating fish ≥4 times per week.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2013-01-09 (Actual); Primary Completion 2017-05-11 (Actual); Study Completion 2017-11-11 (Actual)

PRIMARY OUTCOMES:
Total score of the Hamilton Rating Scale for Depression(HAMD) | Twelve weeks
  The Hamilton Rating Scale for Depression (HAMD) is a commonly used clinical tool for assessing the severity of depression. The most frequently used version, the HAMD-17, includes 17 items and has a total score range from 0 to 52. Higher scores indicate more severe depressive symptoms and thus a worse outcome, while lower scores suggest milder symptoms or improvement.

SECONDARY OUTCOMES:
Total score of the Hamilton Rating Scale for Depression(HAMD) | 4-6 weeks after childbirth
  The Hamilton Rating Scale for Depression (HAMD) is a commonly used clinical tool for assessing the severity of depression. The most frequently used version, the HAMD-17, includes 17 items and has a total score range from 0 to 52. Higher scores indicate more severe depressive symptoms and thus a worse outcome, while lower scores suggest milder symptoms or improvement.
Total scores on the Edinburgh Postnatal Depression Scale(EPDS) | Twelve weeks, 4-6 weeks after childbirth
  The Edinburgh Postnatal Depression Scale (EPDS) is a screening tool used to identify symptoms of postpartum depression. It consists of 10 items, each scored from 0 to 3, giving a minimum total score of 0 and a maximum total score of 30. Higher scores indicate more severe depressive symptoms, meaning a worse outcome, while lower scores suggest fewer or milder symptoms.
Total score of the Beck Depression Inventory II (BDI-II) | Twelve weeks, 4-6 weeks after childbirth
  The Beck Depression Inventory-II (BDI-II) is a widely used self-report questionnaire designed to assess the severity of depressive symptoms. It includes 21 items, each scored from 0 to 3, resulting in a minimum total score of 0 and a maximum total score of 63. Higher scores indicate more severe depression, meaning a worse outcome, while lower scores reflect fewer or less severe symptoms.
Major depressive disorder(MDD)as determined by the depression module of the Mini International Neuropsychiatric Interview (MINI) | Twelve weeks, 4-6 weeks after childbirth
Omega-3 fatty acids concentrations in erythrocytes | Twelve weeks, 4-6 weeks after childbirth
Brain-derived neurotrophic factor(BDNF)in serum | Twelve weeks, 4-6 weeks after childbirth
Estrogen in serum | Twelve weeks, 4-6 weeks after childbirth
Oxytocin in serum | Twelve weeks, 4-6 weeks after childbirth
Progesterone in serum | Twelve weeks, 4-6 weeks after childbirth
Human chorionic gonadotropin (hCG)in serum | Twelve weeks, 4-6 weeks after childbirth
Phospholipase A2 in plasma | twelve weeks, 4-6 weeks after childbirth

OTHER OUTCOMES:
Gestational age | 1 month after childbirth
Gestational diabetes mellitus | 1 month after childbirth
Gestational hypertension or preeclampsia | 1 month after childbirth
Induced labor | 1 month after childbirth
Estimated blood loss | 1 month after childbirth
Cesarean section | 1 month after childbirth
Operative vaginal delivery | 1 month after childbirth
Birthweight | 1 month after childbirth
1-min and 5-min Apgar scores | 1 month after childbirth

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo Medicial University, Shinjuku-Ku, Tokyo, Japan